CLINICAL TRIAL: NCT00216437
Title: A Phase I Dose Escalation Study to Assess the Maximum Tolerated Dose and Feasibility of Combining Oral Capecitabine (Xeloda) and Conformal Radiotherapy (CRT) for Patients With Unresectable Hepatocellular Carcinoma, Multiple Hepatic Metastases or Cholangiocarcinoma
Brief Title: Dose Escalation Study Combining Oral Capecitabine (Xeloda) and Radiotherapy for Patients With Unresectable Liver or Cholangiocarcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: James A. Haley Veterans Administration Hospital (U.S. Federal Agency)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XEL346
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2007-11-12 (Estimated); Status verified 2007-11

CONDITIONS: Cancer of Liver
Keywords: Liver cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Capecitabine

INTERVENTIONS:
Drug: Capecitabine (Xeloda)

SUMMARY:
Our long-term working hypothesis is that if 3-D radiation is combined with the effect of capecitabine one hopes to see improved and durable tumor response and survival with acceptable toxicity. The primary objective is to determine the maximum tolerated dose of capecitabine used along with 3-D conformal radiation therapy.

Capecitabine will be taken by mouth each day of radiation. The total daily dose should be taken as two divided doses approximately 12 hours apart, within 30 minutes after eating, ideally after breakfast and the evening meal. The overall total number of patients expected to participate in this study could be as high as 30 depending on how the treatment is tolerated.

The first group (3-6 patients) on the study will receive the drug (Xeloda®) at 600mg/m² (level 1) and radiation. If the first group does well, the second group of patients on the study (3-6 patients) will receive 825 mg/m² (level 2) and radiation. If the second group does well, the third group will receive 1,000 mg/m² (level 3) and radiation. If the first dose level of 600mg/m² is NOT tolerated, we will reduce the dose to 500mg/m² and enroll another 3-6 patients at the lower dose.

After the highest tolerated dose is identified, 12 additional patients will be treated at that dose to further test the safety of the treatment and better understand the effects of the treatment on disease with more patients.

The following tests and procedures are part of regular medical treatment (standard care) for the disease and are also required for this study.

* physical examinations
* blood tests including pregnancy test
* urinalysis
* ECG (heart tracing)
* chest X-ray
* CT scan of the abdomen

Follow-up visits are done 1 month after radiation, then 3 months later, then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
* Age >18 years
* Ambulatory outpatients (if applicable), with Karnofsky performance status of >60
* Histologically or cytologically confirmed unresectable hepatocellular carcinoma, liver mets with no evidence of extrahepatic disease, or cholangiocarcinoma. (see exclusion criteria 10)
* At least one measurable lesion according to the RECIST criteria which has not been irradiated (i.e. newly arising lesions in previously irradiated areas are accepted). Ascites, pleural effusion, and bone metastases are not considered measurable. Minimum indicator lesion size: > 10 mm measured by spiral CT or >20mm measured by conventional techniques.
* Protocol Specific Laboratory Values as described below in section 6.9 number15.
* Has a negative serum pregnancy test within 7 days prior to start of therapy (female patients of childbearing potential).
* Have concomitant medications been reviewed with patient to address contraindicated medications described in protocol section 6.2.8 and have precautions been taken as recommended for each drug? Includes Allopurinol, Cimetidine, Sorivudine and Brivudine, Anticoagulants, Phenytoin, and Laxatives.

Exclusion Criteria:

* Pregnant or lactating woman. Woman of childbearing potential with either a positive or no pregnancy test at baseline. Woman or men of childbearing potential not using a reliable and appropriate contraceptive method. (Postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential). Patients will agree to continue contraception for 30 days from the date of the last study drug administration
* Life expectancy < 3 months.
* Serious, uncontrolled, concurrent infection(s).
* Any prior fluoropyrimidine therapy (unless given in an adjuvant setting and completed at least 12 months earlier).
* Prior unanticipated severe reaction to fluoropyrimidine therapy, known sensitivity to 5-fluorouracil or known DPD deficiency.
* Completion of previous chemotherapy regimen < four weeks prior to the start of study treatment, or with related toxicities unresolved prior to the start of study treatment.
* Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer.
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
* Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
* Evidence of extrahepatic disease or history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake
* Other serious uncontrolled medical conditions that the investigator feels might compromise study participation.
* Major surgery within 4 weeks of the start of study treatment, without complete recovery.
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
* Known, existing uncontrolled coagulopathy
* Any of the following laboratory values:

  * Abnormal hematologic values (neutrophils < 1.5 x 109/L, platelet count < 100 x 109/L)
  * Impaired renal function (estimated creatinine clearance <50ml/min as calculated with Cockroft-Gault equation.
  * Serum bilirubin > 2.0 x upper normal limit.
  * AST, ALT (SGOT/SGPT) > 2.5 x upper normal limit (or > 5 x upper normal limit in the case of liver metastases).
  * Alkaline phosphatase > 2.5 x upper normal limit (or > 5 x upper normal limit in the case of liver metastases).
* Unwillingness to give written informed consent or provide HIPAA privacy authorization.
* Unwillingness to participate or inability to comply with the protocol for the duration of the study.
* Patient taking a contraindicated medication(s) described in section 6.2.8 (see inclusion criteria #8 for list of agents) and no appropriate substitute agent is available, or patient unable or refuses to take substitute agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-12; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Kazem, MD, Principal Investigator — James A. Haley Veterans Administration Hospital
Locations (1):
- James A. Haley Veterans Administration Hospital, Tampa, Florida, United States